CLINICAL TRIAL: NCT01568996
Title: A Pilot Study Evaluation of Sulforaphane in Atypical Nevi--Precursor Lesions: Assessment of STAT1 and STAT3 Risk Markers of Melanoma
Brief Title: Pilot Study Evaluating Sulforaphane in Atypical Nevi-Precursor Lesions
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: John Kirkwood (Other)
Responsible Party: Sponsor-Investigator, John Kirkwood, Professor and Vice Chairman for Clinical Research, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-114; 10-114 (Other: University of Pittsburgh Cancer Institute (UPCI))
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Atypical Nevi; Melanoma
Keywords: atypical nevi; melanoma; sulforaphane; broccoli; lesions; STAT1; STAT3
MeSH Terms: conditions — Dysplastic Nevus Syndrome; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose BSE-SFN (Experimental): BSE-SFN will be orally administered at 50 µmol SFN for 28 days.
  Interventions: Drug: broccoli sprout extract - sulforaphane (BSE-SFN)
- Mid dose BSE-SFN (Experimental): BSE-SFN will be orally administered at 100 µmol SFN for 28 days.
  Interventions: Drug: broccoli sprout extract - sulforaphane (BSE-SFN)
- High dose BSE-SFN (Experimental): BSE-SFN will be orally administered at 200 µmol SFN for 28 days.
  Interventions: Drug: broccoli sprout extract - sulforaphane (BSE-SFN)

INTERVENTIONS:
Drug: broccoli sprout extract - sulforaphane (BSE-SFN) — 50 µmol capsules, taken orally, once a day for 28 days
  Arms: Low dose BSE-SFN
Drug: broccoli sprout extract - sulforaphane (BSE-SFN) — 100 µmol capsules, taken orally, once a day for 28 days
  Arms: Mid dose BSE-SFN
Drug: broccoli sprout extract - sulforaphane (BSE-SFN) — 200 µmol capsules, taken orally, once a day for 28 days
  Arms: High dose BSE-SFN

SUMMARY:
This is a pilot study to see if oral administration of freeze dried, powdered broccoli sprouts have any effect on whether moles end up becoming melanoma.

DETAILED DESCRIPTION:
This study is designed as a pilot evaluation of sulforaphane as a candidate natural nutritional chemopreventive agent able to modulate key steps in melanoma progression and the expression of STAT proteins in melanocytic and stromal elements of atypical nevi, which are precursor lesions and risk markers of melanoma. Eighteen individuals in total will receive oral broccoli sprout extract rich in sulforaphane (BSE-SFN) standardized for 3 different concentrations of actual sulforaphane content which will be utilized in our study. Three groups of six patients will be randomly assigned to receive oral BSE-SFN at SFN dosages of 50 µmol, 100 µmol, or 200 µmol daily. Due to the established safety of SFN at all of the proposed dosage levels, there is no plan to complete a lower dosage level prior to escalating to the next higher dosage level; i.e., subjects will be randomized across all of the proposed SFN dosage levels. However, the safety of BSE-SFN administration will continue to be evaluated through laboratory studies (CBC, chemistry) performed before and following 28 days of administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have at least two atypical nevi of ≥ 4 mm diameter and prior diagnosis of melanoma.
* Subjects must be ≥ age 18.
* Subjects must not have received any form of systemic antineoplastic treatment for melanoma within the last year from day 1.
* Subjects should not have known allergies to cruciferous vegetables.
* Subjects must agree to abstain from dietary sources of glucosinolates and isothiocyanates beginning three days prior to study and throughout duration of the active study (28 days). Participants will be asked to keep a food diary. A list of food and supplements to abstain from is provided in Appendix A. Patients will be asked to record instances of accidental ingestion of these foods, with patients being removed from the study if this occurs 7 or more times.
* Female subjects must not be pregnant or breast feeding within 6 months prior to and during course of study.
* CBC including diff & platelets - without clinically significant abnormalities
* CMP (Na, K, Cl, CO2, glucose, BUN, creatinine, calcium, total protein, albumin, AST, ALT, ALK phos, total bilirubin) - within 2x ULN

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Adverse events associated with oral sulforaphane | 2 years
Visual changes of atypical nevi: size, border, color. | 2 years
Cellular changes of the atypical nevi. | 2 years

SECONDARY OUTCOMES:
Sulforaphane levels in the blood as a result of the 3 doses. | 2 years
Effects of sulforaphane on STAT1 and STAT3 expression. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John M Kirkwood, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States